CLINICAL TRIAL: NCT01044030
Title: Xylitol Syrup for the Prevention of Acute Otitis Media in Otitis-prone Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Louis Vernacchio, Principal Investigator, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 09-09-0455; RC1DC010668-01 (NIH)
Record Dates: First submitted 2010-01-06; First posted 2010-01-07 (Estimated); Results first posted 2015-03-20 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-05

CONDITIONS: Acute Otitis Media
Keywords: otitis media; ear infection
MeSH Terms: conditions — Otitis Media; Otitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Xylitol syrup (Experimental)
  Interventions: Drug: Xylitol syrup
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Xylitol syrup — 7.5 mL (5 grams) by mouth three times daily
  Arms: Xylitol syrup
Drug: Placebo — 7.5 mL by mouth three times daily
  Arms: Placebo

SUMMARY:
The primary objective of the proposed study is to determine the effectiveness and safety of orally administered viscous-adherent xylitol syrup given in a dose of five grams three times daily for 12 weeks in reducing the incidence of clinically-diagnosed acute otitis media (ear infection) in children with a history of recurrent acute otitis media.

ELIGIBILITY:
Inclusion Criteria:

* Six months to five years of age
* General good health
* History of at least three episodes of AOM in previous 12 months, at least one of which occurred within the previous six months
* English or Spanish speaking

Exclusion Criteria:

* History of tympanostomy tubes
* Intestinal malabsorption or chronic diarrhea
* Diabetes mellitus
* Any inborn error of metabolism
* Parent/guardian unreachable by telephone
* Known allergy to any of the study solution components (xylitol, sorbitol, sodium carboxymethylcellulose, potato starch, glycerin, potassium sorbate, natural berry flavoring).

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 326 (Actual)
Dates: Start 2010-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louis Vernacchio, MD, MSc, Principal Investigator — Boston Children's Hospital
Locations (2):
- United States (2):
  - Children's Hospital Boston, Boston, Massachusetts
  - Slone Epidemiology Center at Boston University, Boston, Massachusetts

REFERENCES:
- [Background] Vernacchio L, Vezina RM, Mitchell AA. Tolerability of oral xylitol solution in young children: implications for otitis media prophylaxis. Int J Pediatr Otorhinolaryngol. 2007 Jan;71(1):89-94. doi: 10.1016/j.ijporl.2006.09.008. Epub 2006 Nov 9. PMID 17097152
- [Result] Vernacchio L, Corwin MJ, Vezina RM, Pelton SI, Feldman HA, Coyne-Beasley T, Mitchell AA. Xylitol syrup for the prevention of acute otitis media. Pediatrics. 2014 Feb;133(2):289-95. doi: 10.1542/peds.2013-2373. Epub 2014 Jan 6. PMID 24394686

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Xylitol Syrup | Placebo
Started | 160 | 166
Completed | 141 | 146
Not Completed | 19 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Xylitol Syrup | Placebo | Total
Number analyzed (Participants) | 160 | 166 | 326
Age, Continuous [Mean (Standard Deviation); unit: months] | 22.3 (13.7) | 21.5 (13.7) | 21.9 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 73 | 140
  Male | 93 | 93 | 186
Race/Ethnicity, Customized [Number; unit: participants]
  White, non-Hispanic | 110 | 114 | 224
  Hispanic | 25 | 22 | 47
  Black, non-Hispanic | 7 | 8 | 15
  Other/Refused/unknown | 18 | 22 | 40

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of Viscous-adherent Xylitol Syrup in Reducing Episodes of Clinically-diagnosed Acute Otitis Media
Description: Proportion of subjects who remained free of acute otitis media throughout the study period
Time Frame: 12 weeks
Measure: Number; unit: percentage of particpants
Arm/Group | Xylitol Syrup | Placebo
Number analyzed (Participants) | 160 | 166
percentage of particpants | 66.9 | 63.3
Statistical Analysis 1: Comparison: Xylitol Syrup vs Placebo; Test type: Superiority or Other; p = 0.6, Chi-squared

2. Secondary Outcome: Effectiveness of Viscous-adherent Xylitol in Reducing Antibiotic Use in Children With Recurrent Acute Otitis Media
Description: Proportion of subjects with no antibiotic use during the study period
Time Frame: 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Xylitol Syrup | Placebo
Number analyzed (Participants) | 160 | 166
percentage of participants | 60.6 | 56.0

3. Secondary Outcome: Effect of Viscous-adherent Xylitol on Nasopharyngeal and Oropharyngeal Colonization With Streptococcus Pneumoniae and Nontypeable Haemophilus Influenzae
Description: Proportion of subjects acquiring colonization with Streptococcus pneumoniae and/or nontypeable Haemophilus influenzae among the subset of patients recruited at the local enrolling sites
Time Frame: 12 weeks
Population: This outcome measure is limited to those subjects enrolled in the local enrolling sites only.
Measure: Number; unit: percentage of participants
Arm/Group | Xylitol Syrup | Placebo
Number analyzed (Participants) | 23 | 20
percentage of participants | 30.4 | 20.0

4. Secondary Outcome: Antimicrobial Resistance Patterns of Isolates of Streptococcus Pneumoniae and Nontypeable Haemophilus Influenzae Cultured From the Oropharynx and/or Nasopharynx of Subjects Treated With Viscous-adherent Xylitol Compared to Placebo.
Description: Proportion of subjects colonized with antibiotic resistant S. pneumonia after treatment
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Xylitol Syrup | Placebo
Number analyzed (Participants) | 17 | 14
Participants
  Resistant | 5 | 6
  Sensitive | 12 | 8

5. Secondary Outcome: Antimicrobial Resistance Patterns of Isolates of Streptococcus Pneumoniae and Nontypeable Haemophilus Influenzae Cultured From the Oropharynx and/or Nasopharynx of Subjects Treated With Viscous-adherent Xylitol Compared to Placebo.
Description: Proportion of subjects colonized with antibiotic resistant nontypeable H. influenzae after treatment
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Xylitol Syrup | Placebo
Number analyzed (Participants) | 16 | 17
Participants
  Resistant | 10 | 7
  Sensitive | 6 | 10

ADVERSE EVENTS:
Arm/Group | Xylitol Syrup | Placebo
Serious Adverse Events (participants affected / at risk) | 4/160 | 1/166
Other Adverse Events (participants affected / at risk) | 89/160 | 93/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Xylitol Syrup (N=160) | Placebo (N=166)
Tympanostomy tube insertion and adenoidectomy (Ear and labyrinth disorders) | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 1 | 0
Abscess (Skin and subcutaneous tissue disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Xylitol Syrup (N=160) | Placebo (N=166)
Diarrhea (Gastrointestinal disorders) | 80 | 84
Flatulence (Gastrointestinal disorders) | 32 | 35
Abdominal Pain (Gastrointestinal disorders) | 15 | 8
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 63 | 58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No